CLINICAL TRIAL: NCT04204070
Title: Comparing Between Ultrasound Assisted Epidural Catheter Placement Using Accuro and the Use of Ultra Sound Real Time With Acoustic Puncture Assisted Device to Confirm Epidural Space End Point
Brief Title: Accuro and the Use of Real Time Ultra Sound With Acoustic Puncture Assisted Device to Confirm Epidural Space End Point
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Yasser Mohamed Mohamed Osman, assistant professor of anesthesia Alexandria university, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 134/200
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Two Different Techniques to Perform Epidural Using Ultrasound
MeSH Terms: interventions — 3-acetylpyridine adenine dinucleotide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I Accuro (Experimental): epidural catheter insertion using the Accuro ultrasound imaging assisted technique
  Interventions: Procedure: Accuro
- Group II APAD (Experimental): epidural catheter insertion using the real time ultrasound guided technique combined with the use of the acoustic puncture assist device (APAD) technique.
  Interventions: Procedure: APAD

INTERVENTIONS:
Procedure: Accuro — A research coordinator recorded the depth of the EDS from skin, the number of attempts to perform the epidural anesthesia, the repositioning of the epidural needle either in the same space or in different space, the time taken for space localisation (it is defined as time taken in seconds from skin puncture until the successful space localisation).the total time of the procedure ( time measured from the patient is fully draped and in the proper sitting position till the end of insertion of the epidural catheter ) Any complications such as paresthesia during catheter insertion, dural puncture, blood in catheter and root irritation will be recorded
  Arms: Group I Accuro
Procedure: APAD — APAD
  Arms: Group II APAD

SUMMARY:
Aim of the work:

To compare the use of the Accuro ultrasound and a real time ultrasound guided epidural combined with the acoustic puncture assisted device to perform the epidural anesthesia Secondary aim is to compare the incidence of complications associated with each technique.

Patient's selection:

This study will be performed on 100 pregnant patients scheduled for normal vaginal delivery under epidural analgesia.

The sample size was calculated by taking success rate of conventional LOR to be 98% in the patients; assuming 80% power, with 95% confidence interval (CI) of two techniques and 30% margin of error.

The study protocol will be reviewed and approved by the Ethics Committee of the Alexandria Main University Hospitals.

A written consent will be obtained from all the patients participating in this study.

Complete history will be taken from all the patients and will be subjected to thorough examination and routine laboratory investigations. Patients will be randomly divided into two equal groups using a computer-generated program.

Group I consists of 50 patients scheduled for epidural catheter insertion using the Accuro ultrasound imaging assisted technique.

Group II consists of 50 patients scheduled for epidural catheter insertion using the real time ultrasound guided technique combined with the use of the acoustic puncture assist device (APAD) technique.

ELIGIBILITY:
Inclusion Criteria:

* pregnant patients scheduled for normal vaginal delivery under epidural analgesia.

Exclusion Criteria:

* • Any contraindication for epidural analgesia

  * High risk pregnancy or precious baby.
  * Patients not willing for participation.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 100 (Estimated)
Dates: Start 2019-08-11 (Actual); Primary Completion 2020-06-11 (Estimated); Study Completion 2020-06-11 (Estimated)

PRIMARY OUTCOMES:
the depth of the EDS from skin, | the procedure time
  inmm
the number of attempts to perform the epidural anesthesia, the repositioning of the epidural needle either in the same space or in different space | the procedure time
  the number of attempts to perform the epidural anesthesia, the repositioning of the epidural needle either in the same space or in different space
, the time taken for space localisation . | the procedure time
  (it is defined as time taken in seconds from skin puncture until the successful space localisation)
the total time of the procedure | the procedure time
  ( time measured from the patient is fully draped and in the proper sitting position till the end of insertion of the epidural catheter )

SECONDARY OUTCOMES:
compare the incidence of complications associated with each technique. | the procedure time
  compare the incidence of complications associated with each technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP